

SEDE LEGALE: Corso Bramante, 88/90 - 10126 Torino Centralino: tel. +39.011.6331633 P.I./Cod. Fisc. 10771180014 www.cittadellasalute.to.it

Presidi Ospedalieri: - Molinette, Dermatologico S. Lazzaro, S. Giovanni Antica Sede - centr. tel. +39.0116331633

- Centro Traumatologico Ortopedico, Istituto Chirurgico Ortopedico Regina Maria Adelaide - centr. tel. +39.0116933111

- Infantile Regina Margherita, Ostetrico Ginecologico S. Anna - centr. tel. +39.0113134444

*Official Title:* Comparing the Efficacy of Dietary Strategies in Managing Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): a Randomized Controlled Trial.

**Document upload:** Informed Consent Form

Document date: Version1.0 August 20,2021.

NCT number: Not available



**SEDE LEGALE:** Corso Bramante, 88/90 - 10126 Torino **Centralino:** tel. +39.011.6331633 **P.I./Cod. Fisc.** 10771180014

www.cittadellasalute.to.it

Presidi Ospedalieri: - Molinette, Dermatologico S. Lazzaro, S. Giovanni Antica Sede - centr. tel. +39.0116331633

- Centro Traumatologico Ortopedico, Istituto Chirurgico Ortopedico Regina Maria Adelaide - centr. tel. +39.0116933111

- Infantile Regina Margherita, Ostetrico Ginecologico S. Anna - centr. tel. +39.0113134444

## INFORMED CONSENT FORM

Title: Comparing the Efficacy of Dietary Strategies in Managing Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): a Randomized Controlled Trial.

Version 1.0, August 20, 2021. **Protocol Code:** Dieta\_NAFLD Sponsor: Department of Medical Sciences, University of Torino **Sponsor Contact:** Prof. Simona Bo **Investigative Site:** Gastroenterology Unit, A.O.U. Città della Salute e della Scienza di Torino **Principal Investigator:** Prof. Elisabetta Bugianesi Email: elisabetta.bugianesi@unito.it — Tel. 011-633 3532 I, the undersigned on **Participant's Statement** I have received detailed and comprehensible explanations regarding the proposed study. I have read and understood all the information contained in the information sheet. I have had the opportunity to speak with the physician and to ask all the necessary questions. I am satisfied with the answers I have received. I have had sufficient time to consider the invitation and make my decision. I understand that I may withdraw my consent at any time (either verbally or in writing), without providing any justification and without any impact on my usual medical care. I have received a copy of the study information sheet, the informed consent form, and the information and consent form regarding the processing of personal data. The originals are kept at the study center. I have received the information sheet to be transmitted to my primary care physician. I hereby voluntarily agree to participate in the above-mentioned study. I consent to the collection of biological samples for the purposes and according to the procedures described in the study. Date Participant's signature Date Signature of the physician providing information

Signature of the participant's legal representative/guardian

(only in case of patient's inability)

Date